CLINICAL TRIAL: NCT06510881
Title: Single Stage Versus Multiple Staged Repair of Nasal & Alveolar Deformities in Patients With Cleft Lip and Palate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youssef Saleh, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Post cleft rhinoplasty
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cleft Lip and Palate; Rhinoplasty
MeSH Terms: conditions — Cleft Lip | interventions — Rhinoplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients at or above age of 8 years for combined rhinoplasty and alveolar repair
  Interventions: Procedure: Rhinoplasty with or without cleft alveolus repair
- Group B (Experimental): patients below 8 years for rhinoplasty alone and a planned alveolar repair in an upcoming session before canine eruption .
  Interventions: Procedure: Rhinoplasty with or without cleft alveolus repair

INTERVENTIONS:
Procedure: Rhinoplasty with or without cleft alveolus repair — * Group (A) : Correction of nasal deformity will be carried out using costochondral cartilage strut for support of septum and lengthening of columella . A concomitant iliac bone graft is taken to reconstruct the alveolar bone . This group age will be above 8 years .
  * Group (B) : Patients who present early before age of 8 years will have rhinoplasty session only . Another session will be prepared for cleft alveolus at age of 8 years .

SUMMARY:
Cleft lip and palate patients are commonly seen among maxillofacial patients. Patients with cleft lip and palate have evident cosmetic nasal deformities. The interrupted insertion of orbicularis oris muscle into the columella on the noncleft side forces the premaxilla, columella and caudal nasal septum towards that side. At the same time, as the orbicularis oris inserts into the alar base on the cleft side, the base is pulled laterally, inferiorly and posteriorly. The malformed lower lateral cartilage on the side of the cleft contributes majorly to the deformity of the nasal tip, causing it to be more blunt. A shorter medial crus and longer lateral crus on the cleft side results in a horizontally wider and displaced nostril on the cleft side. In addition, those patients have alveolar bone defect which results in both cosmetic and dental problems. Repair of the deformed nose along with the reconstruction of the alveolar defect may have an advantage over the staged repair in:- decrease the surgical burden on the patient , correction of the facial asymmetry by redeeming the maxillary bony support , peri-alar augmentation and accordingly obtaining faster and better socio-cosmetic benefit .

DETAILED DESCRIPTION:
Patients are assigned randomly into two groups; group (1) for combined rhinoplasty and alveolar repair , and group (2) for alveolar repair alone and a planned rhinoplasty in an upcoming session .

Pre-operative evaluation:

History taking:

Personal history; name, age, gender and occupation . Patient's complaint(s); as dental problems related to cleft alveolus and both cosmetic and obstructive problems related to nasal deformities .

Clinical examination :

Dental assessment and assessment of the nose according to the Final Standardized Cosmesis and Health Nasal Outcomes Survey (SCHNOS criteria) :

1. Having a blocked or obstructed nose
2. Getting air through my nose during exercise
3. Having a congested nose
4. Breathing through my nose during sleep
5. Decreased mood and self-esteem due to my nose
6. The shape of my nasal tip
7. The straightness of my nose
8. The shape of my nose from the side
9. How well my nose suits my face
10. The overall symmetry of my nose

Radiological evaluation:

Computed Tomography (CT) scan of maxillofacial bones .

Laboratory investigations:

Blood picture, coagulation profile, kidney and liver function tests .

Photogrammetric evaluation

Standard facial photographs of the basal view taken before and after operation will be used to evaluate the results. The photos will evaluate : alar base , nasal tip and nasolabial angle .

Operative procedures:

will be carried out by the same team, under general anesthesia, nasotracheal intubation and supine position.

* Group (1) : Correction of nasal deformity will be carried out according to the pattern of deformity and the complaint of the patient as : cartilage strut for septal support and columellar lengthening , repositioning the alar bases or reconstructing the nasal muscular ring . A concomitant iliac bone graft is taken to reconstruct the alveolar bone .
* Group (2) : Patients will have their alveolus repaired . Bone grafting will be done . Another session will be prepared after 6 months for the rhinoplasty session . The same technique regarding iliac bone graft will be done for those patients .

Post-operative :

Patients will be counselled for wound care , oral hygiene and medications as : Antibiotics , analgesics and anti-inflammatory drugs . Functional and cosmetic outcomes will be assessed 6 months postoperatively .

ELIGIBILITY:
Inclusion Criteria:

- Patients with unilateral cleft lip and palate deformities with evident nasal and cleft lip and palate aged between 5 - 18 years.

Exclusion Criteria:

* * Patients with bilateral complete cleft palate .

  * Patients with only cleft lip.
  * Patients with cleft secondary palate.
  * Patients non fit for surgery.
  * Patients refuse the consent.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of SCHNOS criteria in both groups for evaluation of both cosmetic and functional improvement . The patients will be assessed on the scale and compared between the obtained pre and post operative results after 6 months of surgery . | 6 months after surgery
  1. Having a blocked or obstructed nose
  2. Getting air through my nose during exercise
  3. Having a congested nose
  4. Breathing through my nose during sleep
  5. Decreased mood and self-esteem due to my nose
  6. The shape of my nasal tip
  7. The straightness of my nose
  8. The shape of my nose from the side
  9. How well my nose suits my face
  10. The overall symmetry of my nose

CONTACTS AND LOCATIONS:
Overall Officials: Salaheldin Shaltout, MD, Study Chair — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] DeVictor SR, Tollefson TT. Rhinoplasty in Patients with Cleft Lip Nasal Deformity: Correcting the Alar Base. Facial Plast Surg. 2023 Dec;39(6):668-673. doi: 10.1055/a-2127-3665. Epub 2023 Jul 11. PMID 37433309
- [Result] Phillips S, Hauc SC, Sasson DC, Khetpal S, Ihnat JM, Boroumand S, Rodriguez J, Prassinos A, Lopez J, Steinbacher DM. Sociodemographic Disparities in Access to Cleft Rhinoplasty. J Craniofac Surg. 2023 Jan-Feb 01;34(1):92-95. doi: 10.1097/SCS.0000000000008908. Epub 2022 Aug 17. PMID 35973113
- [Result] Balaji SM. Cleft Rhinoplasty- Columellar lengthening prolabial reconstruction with Abbe flap. Ann Maxillofac Surg. 2016 Jan-Jun;6(1):63-7. doi: 10.4103/2231-0746.186146. PMID 27563610
- [Result] Fisher DM. Unilateral cleft lip repair: an anatomical subunit approximation technique. Plast Reconstr Surg. 2005 Jul;116(1):61-71. doi: 10.1097/01.prs.0000169693.87591.9b. PMID 15988248
- [Result] Patil PG, Nimbalkar-Patil SP. Modified Activation Technique for Nasal Stent of Nasoalveolar Molding Appliance for Columellar Lengthening in Bilateral Cleft Lip/Palate. J Prosthodont. 2018 Jan;27(1):94-97. doi: 10.1111/jopr.12464. Epub 2016 Mar 22. PMID 27002917
- [Result] Liao D, Pereira N, Obayemi A Jr, Sclafani AP. Secondary Cleft Rhinoplasty. Facial Plast Surg Clin North Am. 2024 Feb;32(1):43-54. doi: 10.1016/j.fsc.2023.06.003. Epub 2023 Jul 26. PMID 37981415